CLINICAL TRIAL: NCT02801396
Title: Clinical Evaluation of Investigational Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR-5759
Record Dates: First submitted 2016-05-11; First posted 2016-06-15 (Estimated); Results first posted 2017-06-09 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Visual Acuity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (6):
- Group Sequence A, B, C (Active Comparator): Subjects will wear Test 1, Test 2, and Control contact lenses in order according to the randomization sequence assigned for approximately 30-60 minutes each, with a 5-minute wash-out period between lenses.
  Interventions: Device: Etafilcon A Design 1 (Test 1); Device: Etafilcon A Design 2 (Test 2); Device: Etafilcon A (Control)
- Group Sequence B, C, A (Active Comparator): Subjects will wear Test 1, Test 2, and Control contact lenses in order according to the randomization sequence assigned for approximately 30-60 minutes each, with a 5-minute wash-out period between lenses.
  Interventions: Device: Etafilcon A Design 1 (Test 1); Device: Etafilcon A Design 2 (Test 2); Device: Etafilcon A (Control)
- Group Sequence C, A, B (Active Comparator): Subjects will wear Test 1, Test 2, and Control contact lenses in order according to the randomization sequence assigned for approximately 30-60 minutes each, with a 5-minute wash-out period between lenses.
  Interventions: Device: Etafilcon A Design 1 (Test 1); Device: Etafilcon A Design 2 (Test 2); Device: Etafilcon A (Control)
- Group Sequence C, B, A (Active Comparator): Subjects will wear Test 1, Test 2, and Control contact lenses in order according to the randomization sequence assigned for approximately 30-60 minutes each, with a 5-minute wash-out period between lenses.
  Interventions: Device: Etafilcon A Design 1 (Test 1); Device: Etafilcon A Design 2 (Test 2); Device: Etafilcon A (Control)
- Group Sequence A, C, B (Active Comparator): Subjects will wear Test 1, Test 2, and Control contact lenses in order according to the randomization sequence assigned for approximately 30-60 minutes each, with a 5-minute wash-out period between lenses.
  Interventions: Device: Etafilcon A Design 1 (Test 1); Device: Etafilcon A Design 2 (Test 2); Device: Etafilcon A (Control)
- Group Sequence B, A, C (Active Comparator): Subjects will wear Test 1, Test 2, and Control contact lenses in order according to the randomization sequence assigned for approximately 30-60 minutes each, with a 5-minute wash-out period between lenses.
  Interventions: Device: Etafilcon A Design 1 (Test 1); Device: Etafilcon A Design 2 (Test 2); Device: Etafilcon A (Control)

INTERVENTIONS:
Device: Etafilcon A Design 1 (Test 1)
Device: Etafilcon A Design 2 (Test 2)
Device: Etafilcon A (Control)

SUMMARY:
Single-visit, unmasked, non-dispensing study where subjects will wear three different lenses bilaterally in one visit, each lens being worn for approximately 30-60 minutes. Subjects will complete a questionnaire for each study lens.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be at least 18 years of age and no more than 55 years of age (inclusive).
2. The subject's vertex corrected best spherical distance refraction must be in the range of -1.00 to -6.00 Diopters (D) in each eye.
3. The subject's vertex corrected cylindrical component of distance refraction must be less than or equal to -1.50 Diopters of Cylinder (DC) in each eye.
4. Subjects must have best corrected visual acuity of 20/25 (Snellen or equivalent) or better in each eye.
5. Subjects must self-report as being Asian race.
6. Subjects must self-report as having brown or black eyes.
7. Subjects must be habitual lens wearer (clear or limbal ring cosmetic) . Habitual is defined as at least one (1) month of Contact Lens wear where the lenses were worn for a minimum of six (6) hours per day and a minimum of three (3) days per week.
8. Subjects between 18 to 39 years old must be habitual limbal ring cosmetic lens wearers or must have tried limbal ring cosmetic lens within the past two years.
9. Subjects must be cosmetic contact lens concept acceptors as determined by screening questionnaire.
10. Subjects must possess a functional / usable pair of spectacles and bring them to the visit (only if applicable - to the investigator's discretion).
11. Subjects must read, understand, and sign the Statement of Informed Consent.
12. Subjects must appear able and willing to adhere to the instructions set forth in the clinical protocol.
13. Subjects must be willing to have their eyes video recorded and photographed.

Exclusion Criteria:

1. Working for any advertising agency, any company involved in public relations or marketing, market research; or any company that makes or sells contact lenses or glasses.
2. Participated in any paid market research within the past 3 months.
3. Pregnant or breast feeding a baby.
4. Subjects with diabetes.
5. Any ocular or systemic allergies or disease which might interfere with contact lens wear.
6. Any systemic disease, or autoimmune disease, which might interfere with contact lens wear, at investigator's discretion.
7. Using medications during and immediately preceding the study period that may interfere with current contact lens wear as determined by the investigators
8. Any infectious diseases (e.g. hepatitis, tuberculosis) or a contagious immunosuppressive disease (e.g. HIV), by self-report.
9. Any grade 3 or greater Biomicroscopy findings (this includes, corneal edema, corneal staining, corneal vascularization, conjunctival injection, tarsal abnormalities, bulbar injection) on the FDA classification scale.
10. Any active ocular abnormalities/conditions that might interfere with contact lens wear (this includes, but not limited to, chalazia, recurrent styles, pterygium, infection etc.).
11. Any corneal distortion, scar, or opacity affecting vision as noted by subjects or investigators during examination.
12. History of any corneal surgery (e.g. radial keratotomy (RK), photorefractive keratectomy (PRK), laser-assisted in situ keratomileusis (LASIK)); confirmed with topography if necessary at the investigator's discretion.
13. Habitual wearers of rigid gas permeable or orthokeratology lens within the past 3 months.
14. Current habitual contact lens modality for extended wear or conventional wear (contact lenses with a replacement schedule of 3 months to >1 year).
15. Participation in any pharmaceutical, medical device, or contact lens related clinical research trial within 14 days prior to study enrollment. This excludes studies that do not require product treatment/intervention.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 116 (Actual)
Dates: Start 2016-04-24 (Actual); Primary Completion 2016-05-22 (Actual); Study Completion 2016-05-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hong Kong Polytechnic University, Hong Hom, Kowloon, Hong Kong

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 116 subjects were enrolled into the study. Of the enrolled subjects 15 were not dispensed a study lens. A total of 101 subjects were dispensed a study lens. Of the dispensed subjects 1 was discontinued and 100 subjects completed the study.
Groups:
- Test1/Test2/Control: Subjects that received Test lens 1 during the first period, Test lens 2 during the second period and the Control lens during the third period.
- Test1/Control/Test2: Subjects that received Test lens 1 during the first period, the Control lens during the second period and Test lens 2 during the third period.
- Test2/Test1/Control: Subjects that received Test lens 2 during the first period, Test lens 1 during the second period and the Control lens during the third period.
- Test2/Control/Test1: Subjects that received Test lens 2 during the first period, the Control lens during the second and the Test 1 lens during the third period.
- Control/Test1/Test2: Subjects that received the Control lens during the first period, Test lens 1 during the second period and Test lens 2 during the third period.
- Control/Test2/Test1: Subjects that received the Control lens during the first period, Test 2 lens during the second period and Test lens 1 during the third period.
Period: Period 1
Arm/Group | Test1/Test2/Control | Test1/Control/Test2 | Test2/Test1/Control | Test2/Control/Test1 | Control/Test1/Test2 | Control/Test2/Test1
Started | 17 | 17 | 17 | 16 | 17 | 17
Completed | 17 | 17 | 17 | 16 | 16 | 17
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0
Period: Period 2
Arm/Group | Test1/Test2/Control | Test1/Control/Test2 | Test2/Test1/Control | Test2/Control/Test1 | Control/Test1/Test2 | Control/Test2/Test1
Started | 17 | 17 | 17 | 16 | 16 | 17
Completed | 17 | 17 | 17 | 16 | 16 | 17
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Test1/Test2/Control | Test1/Control/Test2 | Test2/Test1/Control | Test2/Control/Test1 | Control/Test1/Test2 | Control/Test2/Test1
Started | 17 | 17 | 17 | 16 | 16 | 17
Completed | 17 | 17 | 17 | 16 | 16 | 17
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects that were dispensed at least one study lens.
Groups:
- Dispensed Subjects: All subjects that were dispensed at least one study lens.
Arm/Group | Dispensed Subjects
Number analyzed (Participants) | 101
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.43 (9.768)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 45
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 101
Region of Enrollment [Number; unit: Participants]
  China | 101

OUTCOME MEASURES:

1. Primary Outcome: CLUE Handling
Description: CLUE Handling is assessed using the Contact Lens User Experience (CLUE™) Questionnaire. CLUE™ is a validated patient-reported outcomes questionnaire to assess patient experience attributes of soft, disposable contact lenses (comfort, vision, handling, and packaging) in a contact lens-wearing population in the US, ages 18-65. Scores follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable / positive response. 97% of the scores fall within 0 and 120 (mean +/- 3XSD).
Time Frame: 30 Minutes Post Insertion
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Test1: Subjects that wore the Test 1 lens during any of the 3 study periods.
- Test 2: Subjects that wore the Test 2 lens during any of the 3 study periods.
- Control: Subjects that wore the control lens during any of the 3 study periods.
Arm/Group | Test1 | Test 2 | Control
Number analyzed (Participants) | 99 | 99 | 99
Units on a scale | 55.73 (20.146) | 57.58 (20.109) | 64.39 (19.825)

2. Primary Outcome: Visual Performance (LogMar)
Description: Distance time controlled Visual Performance (LogMAR) was assessed for each subject eye under bright-illumination high-contrast lighting conditions at 4m using an ETDRS chart. The average visual performance (LogMAR) was reported for each study lens.
Time Frame: 30 Minutes Post Insertion
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: LogMAR
Units Other Than Participants: Eyes
Arm/Group | Test1 | Test 2 | Control
Number analyzed (Participants) | 99 | 99 | 99
Number analyzed (Eyes) | 198 | 198 | 198
LogMAR | 0.00 (0.082) | 0.00 (0.082) | 0.01 (0.082)

3. Primary Outcome: Percentage of Eyes With Acceptable Mechanical Lens Fit
Description: Mechanical lens fit will be assessed for each subject and eye using a slit lamp. Lens fit is a binary response and 'Yes' = Acceptable Fit and 'No' = Unacceptable Fit. Lens fit is assessed using Lens centration, limbal exposure, primary gaze movement, up-gaze movement, edge lift, lens tightness. Unacceptable fit will be declared if there is any of the following present: limbal exposure, edge lift, excessive movement in primary or up-gaze or insufficient movement in primary gaze and up-gaze. The Percentage of subject eyes with acceptable lens fit will be reported.
Time Frame: 30 Minutes Post Insertion
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Number; unit: Percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Test1 | Test 2 | Control
Number analyzed (Participants) | 99 | 99 | 99
Number analyzed (Eyes) | 198 | 198 | 198
Percentage of eyes | 95 | 97 | 91

4. Primary Outcome: Percentage of Eyes With Acceptable Cosmetic Lens Fit
Description: Cosmetic lens fitting is assessed for each subject eye in the primary gaze position without a slit lamp. Cosmetic lens fit is a binary response and is reported as acceptable or unacceptable. The Percentage of subject eyes with acceptable cosmetic lens fitting is reported.
Time Frame: 30 Minutes Post Insertion
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Number; unit: Percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Test1 | Test 2 | Control
Number analyzed (Participants) | 99 | 99 | 99
Number analyzed (Eyes) | 198 | 198 | 198
Percentage of eyes | 99.5 | 99.5 | 99.5

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study. Approximately 3 hours per subject.
Groups:
- Test2: Subjects that wore the Test 2 lens during any of the 3 periods.
Arm/Group | Test1 | Test2 | Control
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/100 | 0/101
Other Adverse Events (participants affected / at risk) | 0/100 | 0/100 | 0/101

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days